CLINICAL TRIAL: NCT05273827
Title: Clinical Observation of the Effect of Neoadjuvant Anti-PD-1 Immunotherapy on Perioperative Analgesia and Postoperative Delirium in Patients With Non-small Cell Lung Cancer
Brief Title: Effect of Neoadjuvant Anti-PD-1 Immunotherapy on Perioperative Analgesia and Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Tianjin Medical University General Hospital (Other); Tianjin Chest Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2021131
Record Dates: First submitted 2021-10-07; First posted 2022-03-10 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-11

CONDITIONS: Immunotherapy; Analgesia; NSCLC; Delirium
MeSH Terms: conditions — Agnosia; Delirium | interventions — Neoadjuvant Therapy; Paclitaxel; Pemetrexed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be obtained perioperatively. The serum will be further separated and frozen at -80 degrees.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neoadjuvant immunotherapy group: Anti-PD-1 monoclonal antibody (Nivolumab，Pembrolizumab, Sintilimab, or Sugemalimab) 200 mg intravenously in combination with cis-platinum and paclitaxel/pemetrexed
  Interventions: Drug: neoadjuvant immunotherapy
- control group: platinum-containing dual-agent chemotherapy(cis-platinum and paclitaxel/pemetrexed)
  Interventions: Drug: Neoadjuvant chemotherapy

INTERVENTIONS:
Drug: neoadjuvant immunotherapy — Anti-PD-1 antibody was added to the conventional neoadjuvant chemotherapy.
  Other Names: anti-PD-1 therapy
  Groups: neoadjuvant immunotherapy group
Drug: Neoadjuvant chemotherapy — Cis-platinum combined with paclitaxel or pemetrexed
  Other Names: Cis-platinum combined with paclitaxel or pemetrexed
  Groups: control group

SUMMARY:
To observe the effect of preoperative anti-PD-1 monotherapy combined with chemotherapy on patients' perioperative pain and opioid analgesia, and evaluate its effect on the incidence and severity of patients' postoperative delirium.

DETAILED DESCRIPTION:
In this study, the investigators intend to select patients with resectable NSCLC treated with immuno-neoadjuvant therapy in combination with chemotherapy, systematically observe the effect of preoperative anti-PD-1 monotherapy on patients' perioperative pain and opioid analgesia, and evaluate its effect on the incidence and severity of patients' postoperative delirium, in order to provide a clinical basis for the perioperative management of patients treated with immuno-neoadjuvant therapy and promote their postoperative recovery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage II or stage IIIA non-small cell lung cancer (NSCLC) and meet the requirements for R0 resection;
* American Society of Anesthesiologists (ASA): I-III, age ≥18 years, body mass index (BMI): 18.5-30;
* Normal function of Coagulation and vital organs such as heart, lungs, kidney, and liver;
* Eligible to receive platinum-containing two-drug chemotherapy;
* Sign the informed consent form

Exclusion Criteria

* Prior treatment of any kind for current lung cancer, including chemotherapy, radiation or targeted therapy;
* Preoperative opioid analgesia;
* Severe chronic or active infection requiring systemic antibacterial, antifungal or antiviral therapy, including tuberculosis infection;
* History of antipsychotic medication in the last 6 months;
* Preoperative Mini-mental state examination (MMSE) score <23

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NSCLC receiving neo-adjuvant chemotherapy or chemotherapy combined with immunotherapy followed by radical surgery will be screened and recruited in this study.
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
perioperative opioids consumption | from beginning of surgery to day 3 after surgery
  the amount of sufentanil, remifentanil and morphine application.

SECONDARY OUTCOMES:
postoperative delirium | within 3 days after surgery
  record the occurrence of postoperative delirium after surgery using the 3D-CAM test. Patient with postoperative delirium means worse outcome.
score of Numerical Rating Scale | at the time of admission to the operating room, immediately after and at 24 hour, 48 hour, and 72h after entering the PICU
  Record the patient's resting and motor Numerical Rating Scale (NRS) scores, range from 0 to 10, and higher score means more pain.
analgesic pump press in PICU | day 1, 2 and 3 after surgery
  the time of first analgesic pump press and no. of total press in PICU
Percent of patients with moderate to severe pain within 72 hours | up to 72 hours after surgery
  Moderate to severe pain is defined as any NRS pain score of 4 or higher.
intraoperative opioid consumption | from the beginning to the end of the surgery
  the amount of sufentanil and remifentanil
postoperative opioid consumption | up to 72 hours after surgery
  opioid usage in PCIA and supplemental analgesics within 72 h

OTHER OUTCOMES:
dosage of sedatives | intraoperative
  usage of propofol
level of cytokines | before surgery and up to 24 hour after surgery
  IL-6, IL-10, TNF-α, sPD-L1
Pathologic complete response (pCR) rate | up to 30 days after surgery
  0% viable tumor in resected esophagus and lymph nodes
ration of R0 resection | up to 30 days after surgery
  surgical margin is microscopically-negative for residual tumor

CONTACTS AND LOCATIONS:
Overall Officials: Kaiyuan Wang, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (3):
- China (3):
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Tianjin Chest Hospital, Tianjin
  - Tianjin Medical University General Hospital, Tianjin

REFERENCES:
- [Derived] Wang K, Er J, Zhang Y, Song C, Yu Y, Gao R, Xu H, Dong X, Yuan L, Liu Q, Han J, Yu Y, Yin Y. Increased opioid consumption in neoadjuvant immunotherapy plus chemotherapy for patients with non-small-cell lung cancer: A multicenter, prospective cohort study. CNS Neurosci Ther. 2024 Aug;30(8):e14893. doi: 10.1111/cns.14893. PMID 39097916